CLINICAL TRIAL: NCT00972946
Title: The Use of Magnetic Resonance Imaging and Superparamagnetic Particles of Iron Oxide in Cardiovascular Disease - a Pilot Study in Healthy Volunteers
Brief Title: Cell Tracking Using Superparamagnetic Particles of Iron Oxide (SPIO) and Magnetic Resonance Imaging (MRI) - A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Royal College of Surgeons of Edinburgh (Other); Translational Medicine Research Collaboration (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007/R/CAR/15.2
Record Dates: First submitted 2009-09-07; First posted 2009-09-09 (Estimated); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Healthy Volunteer
Keywords: MRI; SPIO

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Administration of labelled cells (Experimental): MRI scanning before and after administration of iron-labelled cells
  Interventions: Biological: Administration of autologous Endorem-labelled mononuclear cells intravenously
- Administration of Endorem (Experimental): MRI scanning before and after intravenous administration of Endorem
  Interventions: Drug: Administration of Endorem

INTERVENTIONS:
Biological: Administration of autologous Endorem-labelled mononuclear cells intravenously — single dose
  Arms: Administration of labelled cells
Drug: Administration of Endorem — single dose, intravenous
  Arms: Administration of Endorem

SUMMARY:
The ability to label specific cells and image their natural movements in vivo would allow researchers to investigate the mechanisms of disease progression. In addition, cell-based therapy, especially stem cell therapy, requires non-invasive monitoring of transplanted cells to follow their bio-distribution and biological function. Because of recent interest in stem cell treatment, several methods have been investigated for in vivo cell tracking. The investigators propose to assess whether the magnetic resonance imaging (MRI) contrast agent Endorem (superparamagnetic particles of iron oxide) can be used to label cells for in vivo tracking using MRI. The investigators will use 20 healthy human volunteers to:

1. Assess the feasibility of imaging Endorem-labelled cells in vivo
2. Compare the distribution of Endorem-labelled cells with that of intravenous injection of Endorem

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age >18 years

Exclusion Criteria:

* Pregnancy
* Contraindication to MRI scanning (detected by safety questionnaire) including severe claustrophobia
* Inability or refusal to give informed consent
* Renal or hepatic dysfunction
* HIV/hepatitis B/ hepatitis C/ HTLV/ syphilis
* Intercurrent illness
* Blood dyscrasias

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2012-01-06 (Actual); Study Completion 2012-01-06 (Actual)

PRIMARY OUTCOMES:
Change in signal intensity in the region of interest on MRI scanning | 0 hours, 24 hours, 48 hours, 5-7 days

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh/Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

REFERENCES:
- [Result] Richards JM, Shaw CA, Lang NN, Williams MC, Semple SI, MacGillivray TJ, Gray C, Crawford JH, Alam SR, Atkinson AP, Forrest EK, Bienek C, Mills NL, Burdess A, Dhaliwal K, Simpson AJ, Wallace WA, Hill AT, Roddie PH, McKillop G, Connolly TA, Feuerstein GZ, Barclay GR, Turner ML, Newby DE. In vivo mononuclear cell tracking using superparamagnetic particles of iron oxide: feasibility and safety in humans. Circ Cardiovasc Imaging. 2012 Jul;5(4):509-17. doi: 10.1161/CIRCIMAGING.112.972596. Epub 2012 Jul 10. PMID 22787016